CLINICAL TRIAL: NCT00503100
Title: Somatosensory Evoked Potentials and Pain Thresholds in Term and Preterm-Born Adolescents After Early Exposure to Pain; a Quantitative Study
Status: Terminated | Type: Observational
Why Stopped: Difficulties in recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Pesach Shvartzman, Head Department of Family Medicine, Soroka University Medical Center
Other Study IDs: SOR458107CTIL
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Somatosensory Disorders
Keywords: Pain; Preterm-Born Adolescents
MeSH Terms: conditions — Somatosensory Disorders; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- NICU full-term early pain group
  Interventions: Device: Thermal stimulation
- NICU premature early pain group
  Interventions: Device: Thermal stimulation
- NICU premature control group
  Interventions: Device: Thermal stimulation
- Soroka- full-term control group
  Interventions: Device: Thermal stimulation

INTERVENTIONS:
Device: Thermal stimulation — Cerebral SEP response (P300, Medoc Ltd., Israel) to thermal stimulation (550C). Warm-sensation threshold (WST), heat-pain threshold (HPT), Cold sensation threshold (CST) and cold pain threshold (CPT) by using Thermal sensory analyzer (TSA-2001,Medoc Ltd., Israel). Pain threshold to tactile stimulation will be measured by using Von-Frey hairs.

SUMMARY:
Background: Several studies have indicated that infants who had undergone postnatal painful procedures appear to be hypersensitive to pain, with a lower threshold to tactile stimulations later on life.

Objective: To study the effect of early exposure to pain on cerebral somatosensory evoked potential (SEP) response to thermal stimulation (550C), in preterm and full term born adolescents (15-18 years old), who have undergone painful procedures during their neonatal period. As well as to study the effect of early exposure to thermal and tactile sensory thresholds and pain thresholds to thermal and tactile stimuli, by using the TSA and von Frey hairs.

Design: Case-control study.

Participants: Four groups of 20 adolescents (aged 15-18 years), two of which are full term and preterm-born who were exposed to painful procedures during the neonatal period. The other two groups are term and preterm-born adolescents who were not exposed to such procedures.

Main Outcome Measures: Cerebral SEP response (P300, Medoc Ltd., Israel) to thermal stimulation (550C). Warm-sensation threshold (WST), heat-pain threshold (HPT), Cold sensation threshold (CST) and cold pain threshold (CPT) by using Thermal sensory analyzer (TSA-2001,Medoc Ltd., Israel). Pain threshold to tactile stimulation will be measured by using Von-Frey hairs.

ELIGIBILITY:
Inclusion Criteria:

For all:

* Age 15-18
* Appropriate weight for gestational age (AGA)
* Informed consent signed by the parent
* Presence of one parent during the examination

Premature groups:

* Preterm-born (32-34 weeks of gestation)
* Admitted to the NICU (ventilated vs. non-ventilated)

Full term groups:

* Completed 37 weeks of gestation Pain groups (premature and full term)
* Admitted to the NICU
* Mechanically-ventilated during the first week of life
* Mechanically-ventilated for at least 48 hours

Exclusion Criteria:

* Current use of analgesia
* A chronic illness with current medical treatment
* Cognitive impairment

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Four groups of 20 adolescents (aged 14 years or older), two of which are full term and preterm-born who were exposed to painful procedures during the neonatal period. The other two groups are term and preterm-born adolescents who were not exposed to such procedures.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cerebral SEP response (P300, Medoc Ltd., Israel) to thermal stimulation (550C). | During the test

SECONDARY OUTCOMES:
Warm-sensation threshold (WST), heat-pain threshold (HPT), Cold sensation threshold (CST) and cold pain threshold (CPT) by using Thermal sensory analyzer (TSA-2001,Medoc Ltd., Israel). | At time of the test
Pain threshold to tactile stimulation will be measured by using Von-Frey hairs | At time of the test

CONTACTS AND LOCATIONS:
Overall Officials: Pesach Shvartzman, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Ben Gurion University of the Negev, Siaal research center for family medicine and primary care, Beersheba, Israel